CLINICAL TRIAL: NCT00756574
Title: A Randomized Control Trial of Surgical Masks vs N95 Respirators to Prevent Influenza in Health Care Workers
Brief Title: Randomized Control Trial to Study the Efficacy of the Surgical Mask Versus the N95 Respirator to Prevent Influenza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6273-15-2008
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2009-08-21 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Influenza
Keywords: N95; Respirator; mask; influenza; efficacy
MeSH Terms: conditions — Influenza, Human | interventions — N95 Respirators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Surgical (Active Comparator): surgical mask
  Interventions: Device: Surgical mask
- 2. N95 Respirator (Active Comparator): N95 respirator
  Interventions: Device: N95 mask

INTERVENTIONS:
Device: Surgical mask — Surgical mask worn for patients with febrile respiratory illness
  Arms: 1. Surgical
Device: N95 mask — N95 mask worn for patients with febrile respiratory illness
  Arms: 2. N95 Respirator

SUMMARY:
The goal of this study is to compare the efficacy of the surgical mask to the N95 respirator in protecting nurses from influenza in the hospital setting. The investigators propose a non-inferiority randomized controlled trial whereby nurses are randomized to either a surgical mask or an N95 respirator when caring for patients with febrile respiratory illness during the influenza season. The hypothesis is that the surgical mask offers similar protection against influenza to that of the N95. The specific objective of the study is to assess whether the rates of influenza (laboratory-confirmed by PCR and HAI assay), as well as secondary outcomes (influenza-like illness, work-related absenteeism, physician visits for respiratory illness, and lower respiratory infection), are similar among nurses using a surgical mask compared to those using an N95 respirator.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who work in emergency departments and medical units
* Nurses expected to work full time (defined as > 37 hours per week)

Exclusion Criteria:

* Nurses who were not fit tested
* Nurses who could not pass a fit test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, MSc, Principal Investigator — Hamilton Health Sciences - McMaster University
Locations (1):
- Hamilton Health Science, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Loeb M, Dafoe N, Mahony J, John M, Sarabia A, Glavin V, Webby R, Smieja M, Earn DJ, Chong S, Webb A, Walter SD. Surgical mask vs N95 respirator for preventing influenza among health care workers: a randomized trial. JAMA. 2009 Nov 4;302(17):1865-71. doi: 10.1001/jama.2009.1466. Epub 2009 Oct 1. PMID 19797474

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1. Surgical | 2. N95 Respirator
Started | 225 | 221
Completed | 212 | 210
Not Completed | 13 | 11
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Surgical | 2. N95 Respirator | Total
Number analyzed (Participants) | 225 | 221 | 446
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 225 | 221 | 446
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (10.6) | 35.8 (10.6) | 36.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 208 | 420
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Canada | 225 | 221 | 446

OUTCOME MEASURES:

1. Primary Outcome: Laboratory-confirmed Influenza Infection
Description: Laboratory confirmed influenza
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | 1. Surgical | 2. N95 Respirator
Number analyzed (Participants) | 212 | 210
participants | 50 | 48

2. Secondary Outcome: Physician Visits for Respiratory Illness
Description: visit to primary care MD
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | 1. Surgical | 2. N95 Respirator
Number analyzed (Participants) | 212 | 210
participants | 13 | 13

3. Secondary Outcome: Influenza-like Illness
Description: Cough and fever
Time Frame: Over entire study period
Measure: Number; unit: participants
Arm/Group | 1. Surgical | 2. N95 Respirator
Number analyzed (Participants) | 212 | 210
participants | 9 | 2

4. Secondary Outcome: Absenteeism
Description: Absent from work because of flu-like illness
Time Frame: over study period
Measure: Number; unit: participants
Arm/Group | 1. Surgical | 2. N95 Respirator
Number analyzed (Participants) | 212 | 210
participants | 42 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No